CLINICAL TRIAL: NCT01206946
Title: Effect of Antenatal Steroids for Women at Risk of Late Preterm Delivery on Neonatal Respiratory Morbidity
Brief Title: Efficacy of Antenatal Steroids in Reducing Respiratory Morbidities in Late Preterm Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Dr. Khalid Yunis, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PED.KY.11
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-09

CONDITIONS: Respiratory Distress Syndrome, Newborn; Transient Tachypnea of the Newborn
Keywords: Respiratory distress; Antenatal steroids; late preterm
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Transient Tachypnea of the Newborn; Dyspnea | interventions — Betamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antenatal steroids (Experimental)
  Interventions: Drug: Betamethasone
- Normal saline (Placebo Comparator)
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Betamethasone — A single course of betamethasone (two doses of 12 mg/dose given at 24 hourly intervals)
  Arms: Antenatal steroids
Other: Normal Saline — Two doses of 2ml of normal saline given at 24 hourly intervals
  Arms: Normal saline

SUMMARY:
The hypothesis of the study is that administration of antenatal steroid to women at high risk of preterm birth after 34 weeks of gestation would reduce the risk of respiratory complications, specifically Respiratory Distress Syndrome (RDS) or Transient Tachypnea of the Newborn (TTN) in late preterm babies.

ELIGIBILITY:
Inclusion Criteria:

* Women between 34 0/7- 36 6/7 weeks of gestation
* High risk of preterm birth

Exclusion Criteria:

* Multiple births
* Fetal congenital malformations
* A course of steroids within 2 weeks of randomization
* Multiple courses of steroids
* Chorioamnionitis
* Non reassuring fetal heart rate
* Obstetrical indication of delivery
* Active bleeding
* Pregnancy related hypertensive disorders
* Uncontrolled diabetes

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory Distress Syndrome (RDS)or Transient Tachypnea of the Newborn(TTN) | First three days of life

SECONDARY OUTCOMES:
Admission to NICU | First three days of life
Hospital stay | Neonatal period (28 days of life)
Days on oxygen | Neonatal period (28 days of life)
Intubations | First three days of life
Surfactant treatment | First three days of life
Pneumothorax | First three days of life
Persistent Pulmonary Hypertension of the Newborn(PPHN) | First three days of life
Days on ventilation | Neonatal period (28 days of life)
Necrotizing enterocolitis (NEC) | Neonatal period (28 days of life)
Clinical sepsis | Neonatal period (28 days of life)
Intraventricular Hemorrhage (IVH) | First week after birth

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Yunis, MD, Principal Investigator — American University of Beirut Medical Center
Locations (5):
- Lebanon (5):
  - American University of Beirut Medical Center, Beirut
  - Bahman Hospital, Beirut
  - Hotel Dieu de France, Beirut
  - Rafik Hariri University Hospital, Beirut
  - St Georges Hospital- University Medical Center, Beirut